CLINICAL TRIAL: NCT06807138
Title: AVF Volume Blood Flow Reduction in HD Patients with Chronic Heart Failure
Brief Title: AVF Volume Blood Flow Reduction in HD Patients
Status: Completed | Type: Observational
Sponsor: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Responsible Party: Principal Investigator, Alexey Zulkarnaev, Leading Researcher, Moscow Regional Research and Clinical Institute (MONIKI)
Other Study IDs: 290125
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease Stage 5; Heart Failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- NYHA I-II: Patients with NYHA I-II heart failure
- NYHA III-IV: Patients with NYHA III-IV heart failure

SUMMARY:
Heart failure with preserved / high cardiac output is a well-known syndrome in patients with high-flow arteriovenous fistula (AVF). However, the threshold for classifying an AVF as high-flow is currently undefined. Cardio-fistular recirculation (CFR) is often used as a criterion, with values greater than 25-30% considered cardiotoxic and associated with adverse outcomes. Additionally, CFR is one of the few easily modifiable risk factors through surgical reduction of AVF volume blood flow (Qa).

The study aimed to evaluate the extent of involution of heart structural and functional changes following Qa reduction in patients with heart failure and CFR > 25%.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* age > 18 years
* CKD 5D
* Native arteriovenous fistula or vascular graft
* Heart failure with preserved CO (NYHA I-IV )
* Cardio-fistula recirculation ≥ 25%
* eKt/V > 1.2
* Absence of arrhythmias (except grade I AV block)
* Absence of valvular disease (except mitral regurgitation I-II)
* Arteriovenous fistula blood flow reduction surgery

Exclusion Criteria:

* Death
* Kidney transplantation
* Conversion of vascular access to central venous catheter
* Withdrawal of informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving maintenance hemodialysis treatment
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | Before and at 6 months after surgery
Estimated pulmonary artery pressure | Before and at 6 months after surgery
E/A ratio | Before and at 6 months after surgery

SECONDARY OUTCOMES:
NT-proBNP serum concentration | Before and at 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow Regional Research and Clinical Institute, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code